CLINICAL TRIAL: NCT03959592
Title: Macular Pigment and Visual Performance in Glaucoma Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Preliminary analysis showed no benefit of the investigational supplement.
Sponsor: Felipe Medeiros, MD (Other)
Collaborators: Heidelberg Engineering GmbH (Industry); MacuHealth (Industry); Industrial Orgánica S.A. de C.V. (Industry)
Responsible Party: Sponsor-Investigator, Felipe Medeiros, MD, Professor of Ophthalmology, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00093041
Record Dates: First submitted 2019-05-17; First posted 2019-05-22 (Actual); Results first posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Lutein; Zeaxanthins

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lutein, zeaxanthin and mesozeaxanthin (Active Comparator): Patients will be asked to consume 1 pill daily with a meal, for six months. The pills will contain 22 mg total of the carotenoids lutein (10 mg), zeaxanthin (2 mg), and mesozeaxanthin (10 mg).
  Interventions: Drug: Lutein, zeaxanthin and mesozeaxanthin
- Placebo (Placebo Comparator): Patients will be asked to consume 1 pill daily with a meal, for six months. The pills will contain only sunflower oil (placebo).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lutein, zeaxanthin and mesozeaxanthin — The intervention will involve supplementation with the macular carotenoids (1 pill daily with a meal containing lutein, zeaxanthin, mesozeaxanthin) for six months, to determine the effects on visual performance in glaucoma patients.
  Other Names: macular carotenoids
  Arms: Lutein, zeaxanthin and mesozeaxanthin
Other: Placebo — This intervention involves an inert pill (1 pill daily with a meal) that contains only sunflower oil, for six months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine cross-sectional relationships between macular pigment optical density (MPOD) and visual performance in glaucoma. Additionally, the investigators wish to determine the effect of lutein, zeaxanthin, and mesozeaxanthin supplementation on MPOD and visual performance in glaucoma patients.

DETAILED DESCRIPTION:
Neurodegeneration of the optic nerve and associated ganglion cell death in glaucoma leads to several well-characterized losses in visual function, most notably progressive peripheral visual field loss. Several recent studies have characterized significant visual function deficits in glaucoma patients that may be more sensitive indicators of disease than classical visual field loss, including compromised contrast sensitivity (CS), increased disability glare (DG) and protracted dark adaptation (DA).

Given the available evidence, it appears that visual function, if assessed carefully, is a reliable indicator of ocular health and/or disease state. It follows that an improvement in visual function would be indicative of an improvement in ocular health. Although improvement of visual function is not typically seen in ocular disease, there is recent evidence to suggest that visual performance and associated progression of ocular disease may actually be modifiable via nutritional strategies and dietary modification in age-related macular degeneration (AMD). Because some of the compromised visual performance experienced in glaucoma is associated with increased ocular inflammation, local anti-inflammatory action may improve visual performance in glaucoma patients. Given their exceptional anti-inflammatory activity and potential for rich deposition in the retina, the macular carotenoids lutein (L), zeaxanthin (Z), and mesozeaxanthin (MZ) may hold promise for this strategy. Indeed, a recent cross-sectional study of the relationship between macular carotenoid level and visual performance in glaucoma patients found that those patients with low levels were significantly more likely to experience problems with glare - and were also more likely to have greater ganglion cell loss.

L and Z are diet-derived, yellow-orange colored carotenoids obtained primarily from leafy-green vegetables. L and Z are not synthesized by the body, and therefore must be obtained via dietary means; those who have diets rich in leafy greens, or supplement with sufficient L and Z tend to maintain and accumulate higher blood and tissue concentrations. One of the conspicuous features of L and Z is their specific accumulation in the macular retina, where they can reach extremely high concentrations - values as high as 1.50 log optical density near the foveal center are not uncommon; it is also not uncommon to see concentrations in the fovea that exceed 10,000 times that seen in the blood. Once deposited in the retina, some of the L is converted to a stereoisomeric form of zeaxanthin, called mesozeaxanthin (MZ). Although rare, MZ has been shown to exist in nature, and indeed in the human food chain - its presence has been recently verified in salmon, trout, and sardine skin, and also trout flesh. Importantly, MZ has been shown to be readily deposited in the retina when taken in supplement form. The accumulation of these three carotenoids in the macula yields a yellowish-orange coloration, classically known to ophthalmologists as the "macula lutea" ("yellow spot"). Today, this collective pigmentation is commonly referred to as macular pigment (MP), with concentrations typically expressed in terms of optical density (MPOD). Xanthophyll carotenoids such as L, Z, and MZ are especially potent antioxidants. Via a process called triplet excitation transfer, L, Z, and MZ can regenerate to repeatedly "quench" the energy of singlet oxygen. This makes them capable of long-term accumulation in target tissues such as the retina, where, in the absence of excessive oxidative or inflammatory stress (e.g. smoking, or systemic disease such as diabetes), they are resistant to turnover, and can provide continuous protection against oxidation and inflammation.

Another critical function of the macular carotenoids involves their optical properties within the eye. Visual discomfort in glare, disability glare, and photostress recovery time are all significantly improved with higher MPOD status. CS has also been found in several laboratories (for both normal and clinical populations) to be related to / enhanced by augmentation of MPOD. Dark adaptation speed, absolute scotopic thresholds, and mesopic contrast sensitivity have also been found to be impacted positively by MPOD.

A high concentration of macular carotenoids (i.e. high MPOD) is therefore advantageous in at least three ways: 1) Protection from oxidation and inflammation, 2) Filtration of potentially actinic high-energy short-wavelength light, and 3) Improvement of visual performance (via pre-receptoral screening of short-wave light and neurophysiological enhancement).

For baseline measures, the proposed study has the potential to determine cross-sectional relationships between MPOD, visual performance, and disease severity in glaucoma. Given the recent data, significant relationships are plausible - and if the investigators determine these kinds of relationships, standard of care for glaucoma patients could be changed to include improved patient education regarding nutrition. Additionally, visual function testing (to include CS, DA, and DG testing) may be instituted for glaucoma suspects and established glaucoma patients. If the investigators are able to show an acute effect of improvement in visual performance, it could lead to larger trials that may yield extremely important data with regard to management of glaucoma. Given the predicted exponential increase in worldwide glaucoma prevalence (76 million in 2020 to 111.8 million in 2040), strategies that may promote good visual function in glaucoma would be hugely significant.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma diagnosis: To be considered glaucomatous, patients will be required to have: (1) history of elevated intraocular pressure (IOP; over 21 mmHg); (2) at least two consecutive and reliable standard automated perimetry (SAP) examinations with either a pattern standard deviation (PSD) outside the 95% normal limits or a glaucoma hemifield test (GHT) result outside the 99% normal limits; and/or glaucomatous optic neuropathy.
* between the ages of 18 and 75 years,
* must be able and willing to provide signed informed consent and follow study instructions.

Exclusion Criteria:

* no systemic disease, no other ocular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe A Medeiros, MD, PhD, Principal Investigator — Duke Eye Center
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lutein, Zeaxanthin and Mesozeaxanthin | Placebo
Started | 3 | 5
Completed | 3 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lutein, Zeaxanthin and Mesozeaxanthin | Placebo | Total
Number analyzed (Participants) | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.9 (3.2) | 61.8 (9.0) | 67.1 (3.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Contrast Sensitivity
Description: Contrast sensitivity is the ability to detect subtle differences in shading and patterns. In temporal contrast sensitivity, a spatially homogeneous disc whose luminance varies sinusoidally over time is presented. Its temporal frequency is measured as the maximum number of cycles in a second (Hz) at which the flickering is perceived by the patient.
Time Frame: Baseline to 6 months
Population: Eyes with low visual acuity were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Hz
Units Other Than Participants: Eyes
Arm/Group | Lutein, Zeaxanthin and Mesozeaxanthin | Placebo
Number analyzed (Participants) | 3 | 5
Number analyzed (Eyes) | 4 | 7
Hz | 3.44 (4.83) | -0.23 (1.90)
Statistical Analysis 1: Comparison: Lutein, Zeaxanthin and Mesozeaxanthin vs Placebo; Test type: Other; p = 0.14, Generalized Estimating Equations

2. Primary Outcome: Change in the Macular Pigment Optical Density
Description: Accumulation of the macular carotenoids (lutein, zeaxanthin, and mesozeaxanthin) occurs in the central retina, and is characterized by its optical density (the ability of the pigment to absorb light). Optical density equals the log to the base 10 of the reciprocal of the transmittance.
Time Frame: Baseline to 6 months
Population: Participants excluded from this analysis if presenting low signal quality due to media opacity.
Measure: Mean (Standard Deviation); unit: Optical density units
Units Other Than Participants: Eyes
Arm/Group | Lutein, Zeaxanthin and Mesozeaxanthin | Placebo
Number analyzed (Participants) | 3 | 2
Number analyzed (Eyes) | 3 | 2
Optical density units | 0.06 (0.06) | 0.02 (0.03)
Statistical Analysis 1: Comparison: Lutein, Zeaxanthin and Mesozeaxanthin vs Placebo; Test type: Other; p = 0.423, Generalized Estimating Equations

3. Secondary Outcome: Change in the Speed of Dark Adaptation
Description: After exposure to a relatively bright environment, visual adaptation to the dark (where one can reliably detect objects in dim light) takes some time.
Time Frame: Baseline to 6 months
Population: Data not collected.
Arm/Group | Lutein, Zeaxanthin and Mesozeaxanthin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Vision in Glare as Measured by Percentage of Contrast
Description: Visual performance, especially contrast sensitivity, is greatly decreased by the presence of glare. Range 0% (white on white) to 100% (black on white) contrast.
Time Frame: Baseline to 6 months
Population: Patients excluded from this analysis if not able to see letter at 100% contrast with glare on in at least one of the visits.
Measure: Number; unit: percentage of contrast
Units Other Than Participants: Eyes
Arm/Group | Lutein, Zeaxanthin and Mesozeaxanthin | Placebo
Number analyzed (Participants) | 1 | 1
Number analyzed (Eyes) | 1 | 1
percentage of contrast | 0 | 48

5. Secondary Outcome: Change in the Quality of Life by the National Eye Institute Visual Function Questionnaire (NEI VFQ-25)
Description: The NEI VFQ-25 is a 25-question visual function quality questionnaire. Values are assigned from 0 to 100 according to the answers to 25 items. Higher values represent a better outcome.
Time Frame: Baseline to 6 months
Population: One subject in the placebo group did not respond to the NEI VFQ-25 at the 6 month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lutein, Zeaxanthin and Mesozeaxanthin | Placebo
Number analyzed (Participants) | 3 | 4
score on a scale | 11.2 (10.8) | 11.0 (14.2)
Statistical Analysis 1: Comparison: Lutein, Zeaxanthin and Mesozeaxanthin vs Placebo; Test type: Other; p = 0.985, Generalized Estimating Equations

6. Secondary Outcome: Change in Visual Field Assessment
Description: A visual field assessment tests the sensitivity of regions across the retina that correspond to points in the visual field. Mean deviation (MD) reflects the overall depression (deviation from normal values) of the field in dB.
Time Frame: Baseline to 6 months
Population: Eyes with visual fields with low reliability score were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: dB
Units Other Than Participants: Eyes
Arm/Group | Lutein, Zeaxanthin and Mesozeaxanthin | Placebo
Number analyzed (Participants) | 3 | 5
Number analyzed (Eyes) | 4 | 7
dB | 0.06 (0.59) | -0.36 (1.65)
Statistical Analysis 1: Comparison: Lutein, Zeaxanthin and Mesozeaxanthin vs Placebo; Test type: Other; p = 0.545, Generalized Estimating Equations

7. Secondary Outcome: Change in the Point-spread Function
Description: The point-spread function describes the optical quality of the eye.
Time Frame: Baseline to 6 months
Population: Data not collected.
Arm/Group | Lutein, Zeaxanthin and Mesozeaxanthin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Lutein, Zeaxanthin and Mesozeaxanthin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT03959592/Prot_SAP_000.pdf